CLINICAL TRIAL: NCT06260618
Title: A Single-blinded Randomised Trial Evaluating the Efficacy of Chitosan-dextran (Chitodex) Gel Versus Gelfoam Sponge Instillation Within the Middle Ear and External Auditory Canal During Tympanoplasty Surgery
Brief Title: Effect of Chitodex Gel in Tympanoplasty Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Adelaide Local Health Network Incorporated (Other Government)
Collaborators: University of Adelaide (Other)
Responsible Party: Principal Investigator, Peter-John Wormald, Prof Peter John Wormald MD, FAHMS, FRACS, FACS, FCS(SA), FRCS (Ed), MBChB Chairman Otolaryngology Head and Neck Surgery Professor of Skull Base Surgery , CAHLN and University of Adelaide, Central Adelaide Local Health Network Incorporated
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/HRE00065
Record Dates: First submitted 2024-01-31; First posted 2024-02-15 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Tympanic Membrane Perforation; Tympanic Membrane Inflammation; Surgery; Otitis Media
Keywords: tympanic membrane; surgery; single blinded; chitogel; chitosan-dextran; otitis media; gelfoam; medical device; chitodex; myringoplasty; mastoidectomy; ossiculoplasty
MeSH Terms: conditions — Tympanic Membrane Perforation; Otitis Media | interventions — Gelatin Sponge, Absorbable

STUDY DESIGN:
Intervention Model Description: Single blinded randomised clinical trial
Who Masked: Participant
Masking Description: Masked: The people receiving the treatment/s, The people analysing the results/data Unmasked: The surgeon administering the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gelfoam Arm (Active Comparator): The current standard of care in middle ear packing material has been Gelfoam, Gelfoam is an absorbable gelatin sponge manufactured from denatured porcine skin. Generally, Gelfoam resides within the middle ear for 2 to 9 weeks prior to being degraded via phagocytosis.
  A single Gelfoam sponge is divided into small pieces and used within the ear. One piece of Gelfoam can typically be cut into over 200 smaller pieces. The surgeon uses approximately 10 to 20 of these smaller pieces per surgery. Approx a third of the product is applied into the middle ear, as a support material for the graft. After graft suturing is complete, the remaining two thirds are applied into the external ear canal as a packing agent.
  The surgeon administers the foam during the surgery as they would with the standard TMP repair surgery. The product comes in a sterile package to be opened and cut up by Scrub Nurse.
  Interventions: Device: Gelfoam
- Chitodex Arm (Experimental): Chitosan-dextran gel is packaged within a syringe and has a cannula attached, much like the Gelfoam syringe system. Approx 3-5mL of product is applied during the surgery. Approx 2mL into the middle ear, as a support material for the graft. After graft suturing is complete, another 3mL (approx) is applied into the external ear canal as a packing agent. This is the same procedure as Gelfoam is currently used for this purpose.
  The surgeon will administer the gel during the surgery as they would with the standard of care Gelfoam. The product comes in a sterile kit to be opened by Scrub Nurse.
  Interventions: Device: Chitodex

INTERVENTIONS:
Device: Gelfoam — GELFOAM Sterile Compressed Sponge is a medical device intended for application to bleeding surfaces as a hemostatic. It is a water-insoluble, off-white, nonelastic, porous, pliable product prepared from purified porcine skin, Gelatin USP Granules and Water for Injection, USP. It may be cut without fraying and is able to absorb and hold within its interstices, many times its weight of blood and other fluids.
  Other Names: Gelfoam® absorbable gelatin compressed sponge, USP
  Arms: Gelfoam Arm
Device: Chitodex — The Chitogel Endoscopic Sinus Surgery Kit contains components and equipment for the preparation of a nasal gel to be applied to the sinus cavities via a supplied and specifically designed malleable cannula.
  The Gel preparation will take approximately 30 minutes, so preparation must start sufficiently in advance of when the Gel is expected to be used in surgery.
  Once the Gel has been prepared it should be applied to the sinus cavities on both sides within six hours using the malleable cannula supplied with the Kit.
  The Gel must be prepared on a sterile surface following these instructions. There are two main components to the Gel.
  1. Dextran Aldehyde (B), which is a dry powder, and is reconstituted into a liquid form through mixing the powder with a liquid Sodium Phosphate Buffer (A). Both of these components are supplied sterile.
  2. The second component Chitosan Succinamide (C), is a liquid and is also supplied sterile.
  Other Names: Chitosan-Dextran, Chitogel Endoscopic Sinus Surgery Kit
  Arms: Chitodex Arm

SUMMARY:
The general purpose of this study is to compare Chitosan-dextran (Chitodex) gel versus current standard of care, Gelfoam, as a middle ear (ME) and external auditory canal (EAC) packing agent as part of tympanoplasty, ossiculoplasty and mastoidectomy procedures.

DETAILED DESCRIPTION:
The general purpose of this study is to compare Chitosan-dextran (Chitodex) gel versus current standard of care, Gelfoam, as a middle ear (ME) and external auditory canal (EAC) packing agent as part of tympanoplasty procedures to close tympanic membrane perforations (TMP), or ossiculoplasty due to ossicular chain disruption and its sequelae, or mastoidectomy for Chromin Otitis Media (COM) or its sequelae eg cholesteatoma.

The investigators aim to compare the success rates of middle ear surgery between the two products. The ultimate goal is to identify the ME packing agent-of-choice to ensure TMP closure as well as minimal inflammation of the middle ear mucosa. The most critical measure of success during tympanoplasty surgery is the closure of a chronic, pre-existing TMP. As such, the primary outcome will be a measure of tympanic membrane closure. This is performed under direct vision during routine post-operative surveillance via the use of either a hand-held otoscope or an operating otologic microscope. The investigators will perform this check at 4 distinct time-points: 2 and 6 weeks post-op, 3 months post-op and 6 months post-op.

Chitosan-dextran gel is packaged within a syringe and has a cannula attached, much like the Gelfoam syringe system. Approx 3-5mL of product is applied during the surgery. Approx 2mL into the middle ear, as a support material for the graft. After graft suturing is complete, another 3mL (approx) is applied into the external ear canal as a packing agent. This is the same procedure as Gelfoam is currently used for this purpose.

The surgeon will administer the gel during the surgery as they would with the standard of care Gelfoam. The product comes in a sterile kit to be opened by Scrub Nurse.

Fidelity of the interventions is measured in several ways by the surgeon at the end of the operation. A good seal for the graft is always assessed for by the surgeon prior to completing any tympanoplasty. This is determined via any evidence of air escape from the middle ear when palpating the tympanic membrane and graft at the end of the procedure. A good seal indicates a well-positioned graft. The surgeon's operative notes will indicate this. The investigators will also obtain endoscopic images and videos at the end of procedure to assess positioning of the graft.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who have otoscopic evidence of tympanic membrane perforation that is also confirmed by tympanometry (Defined as a Type B tympanogram, with elevated EAC volume) AND

   1. The TM perforation is associated with at least 15dB of conductive hearing loss on the affected side AND
   2. Are indicated to undergo closure of the perforation via tympanoplasty surgery
2. OR Individuals who are indicated for ossiculoplasty due to ossicular chain disruption and its sequelae
3. OR Individuals who are indicated for mastoidectomy for COM or its sequelae eg cholesteatoma
4. Demonstrate healthy, dry middle ear mucosal cavities at time of surgery AND
5. Are 18 years of age or over AND
6. Are able to give written informed consent AND
7. Are committed to returning for post-operative assessments at 2 and 6 weeks post-op, 3-, and 6- months post-op

Exclusion Criteria:

1. Operative ear is the better or only hearing ear
2. The ear has evidence of cholesteatoma or other middle ear tumour during otoscopic examination
3. dysfunction during otoscopic and tympanometric examination
4. Known allergy to shellfish or ciprofloxacin antibiotics
5. Pregnant or breastfeeding
6. Hepatitis, HIV or any blood disorders
7. COVID-19 positive patients
8. Contra-indications for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-11-20 (Actual); Primary Completion 2025-05-13 (Estimated); Study Completion 2025-05-13 (Estimated)

PRIMARY OUTCOMES:
Number of participants with tympanic membrane closure | Pre-operatively, and 2 weeks, 6 weeks, 3 months and 6 months post-operatively
  tympanic membrane closure will be assessed via otoscopy (images will be captured via the otoscopic equipment)
rate of tympanic membrane closure | Pre-operatively, and 2 weeks, 6 weeks, 3 months and 6 months post-operatively
  Time taken for tympanic membrane to close, assessed by otoscopy (images will be captured via the otoscopic equipment)

SECONDARY OUTCOMES:
Number of participants with improved hearing | Pre-operatively, and 2 weeks, 6 weeks, 3 months and 6 months post-operatively
  An audiogram will be used for assessment of hearing. It measures hearing thresholds in decibels over a range of noise frequencies from 200Hz up to 8000Hz. It is always performed in a sound-proof room with over ear headphones
Number of participants with improved eardrum function | Pre-operatively, and 3 months and 6 months post-operatively
  Eardrum function will be tested by Tympanometry, which tests how well the eardrum moves. The audiologist will put a small probe into the ear. A small device attached to the probe will push air into the ear. The output from the probe is translated to a graph called a tympanogram.
Ease of use of product compared to active comparator - surgeon feedback | Once, on day of surgery (within 6 hours post-operatively)
  Ease of use of product will be assessed via surgeon's feedback
  The ease of which to place the packing material within the anterior mesotympanum will be assessed, as well as the ease with which adequate graft positioning was obtained at the end of surgery. This will be done on a 7-point Likert scale with 1 been very difficult and 7 being very easy to use. After the surgeon has finished the surgery, the trial staff will collect this score from the surgeon within 24 hours of the surgery.
Time taken to complete surgery | Once, for the duration of the operation (hours)
  Start and finish times for all surgeries is clocked into the hospital peri-operative software by the nursing staff in real time. This is a routine part of modern peri-operative care. These records can be retrieved to establish the total operating time of each surgery.
Number of Participants with improved quality of life | Pre-operatively, and 2 weeks, 6 weeks, 3 months and 6 months post-operatively
  This will be determined by a participant subjective symptom score/questionnaire, called the Modified Chronic Otitis Media Outcomes Test (modCOMOT-8 test).
  This is a modified/shorter version of a validated test that was designed for the current study, as there is no current validated questionnaire to assess post-tympanoplasty subjective symptoms, The original test, The Chronic Otitis Media Outcomes Test (COMOT-15 test) has been published widely.
  The modCOMOT-8 test includes a score for (left and right); hearing, ear discharge, ear pain, ear fullness, tinnitus (ringing in the ears), vertigo, overall ear health, overall impact on quality of life. The total possible score ranges from 0 to 160, where the lower the score, the better the outcome.
Clearance of Chitodex gel from middle ear | 4 weeks post-operatively
  Clearance of Chitodex gel or gelfoam from middle ear will be assessed by Magnetic resonance imaging (MRI). This will determination of clearance the packing agent or of any inflammatory or infectious processes.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Peter-John Wormald, MD, Principal Investigator — Central Adelaide Local Health Network
Locations (2):
- Australia (2):
  - The Queen Elizabeth Hospital, Adelaide, South Australia
  - The Memorial Hospital, North Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No